CLINICAL TRIAL: NCT03982758
Title: Acute Effect of Isometric Physical Exercise on Blood Pressure in Patients With Controlled Hypertension
Brief Title: Acute Effect of Isometric Exercise on Blood Pressure in Hypertensive Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto de Cardiologia do Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Patricia Caetano, principal investigador, Instituto de Cardiologia do Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PCaetano
Record Dates: First submitted 2019-04-15; First posted 2019-06-12 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Arterial Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- isometric handgrip exercise (Experimental): Isometric session with handgrip: 4 sets of 2 minutes of contractions sustained at 30% of CVM, for each arm. The time between sets and between arms will be 1 minute rest.
  Interventions: Other: isometric handgrip exercise
- isometric of lower limbs (Experimental): Isometric session for lower limbs: 4 series with 2 minutes of contractions sustained at 30% of 1RM. The rest interval will be 1 minute.
  Interventions: Other: isometric of the lower limbs

INTERVENTIONS:
Other: isometric handgrip exercise — Isometric session with handgrip: 4 sets of 2 minutes of contractions sustained at 30% of CVM, for each arm. The time between sets and between arms will be 1 minute rest.
  Arms: isometric handgrip exercise
Other: isometric of the lower limbs — Isometric session for lower limbs: 4 sets with 2 minutes of contractions sustained at 30% of 1RM. The rest interval will be 1 minute rest.
  Arms: isometric of lower limbs

SUMMARY:
International recommendations advocate dynamic or isometric strength training as an adjunct to aerobic exercise. Due to a lack of consensus, this research addresses the acute effects of isometric exercises by handgrip or lower limb isometry as a hypotensive strategy in hypertensive adults.

DETAILED DESCRIPTION:
This study is characterized as a randomized, controlled and blinded clinical trial for the evaluators and carried out integrally in the Laboratory of Clinical Investigation (LIC) of the Cardiology Institute of Rio Grande do Sul / University Foundation of Cardiology (ICFUC). The project follows all recommendations proposed by the CONSORT Statement.

The study will consist of individuals of both genders, aged between 40 and 70 years who have blood pressure above 120mmhg by 80mhg. The participants, after signing the informed consent, answered a questionnaire that will evaluate the habitual level of physical activity and will be submitted to isometric exercises of palmar grip or quadriceps muscle. Pre- and post-exercise blood pressure will be monitored through the ambulatory blood pressure monitoring (ABPM) method.

ELIGIBILITY:
Inclusion Criteria:

* Controlled hypertensive patients (use of medication) sedentary or physically inactive

Exclusion Criteria:

* Pregnant women;
* Unstable angina;
* Class II, III or IV heart failure;
* Recent cardiovascular event (last 3 months);
* Chronic renal insufficiency;
* Diabetes;
* History of malignant diseases with life expectancy <2 years;
* Or Orthopedic limitations or any physical or mental limitation that impedes the performance of physical exercises.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-12-09 (Actual); Primary Completion 2022-03-18 (Estimated); Study Completion 2022-03-18 (Estimated)

PRIMARY OUTCOMES:
blood pressure | 48 hours
  Blood pressure will be evaluated by Ambulatory Blood Pressure Monitoring (ABPM) over 24h. For that, a Dyna-Map® branded instrument will be used, which will measure blood pressure on rest condition and another measure after the exercise session (totaling 48 horas), in all participants of the two study groups.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Caetano, graduate, Principal Investigator — Instituto de Cardiologia/ Fundação Universitária de Cardiologia
Locations (1):
- Instituto de Cardiologia/ fundação Universitária de Cardiologia, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Oliveira PC, Dipp T, Waclawovsky G, Lehnen AM. Post-isometric exercise hypotension occurs irrespective of muscle mass in adults with hypertension: A randomized clinical trial. Clinics (Sao Paulo). 2025 Apr 16;80:100612. doi: 10.1016/j.clinsp.2025.100612. eCollection 2025. PMID 40245790